CLINICAL TRIAL: NCT05486897
Title: Periventricular White Matter Hyperintensities in Cerebral Amyloid Angiopathy and Hypertensive Arteriopathy
Acronym: PVWMH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/DR-04
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Amyloid Angiopathy; Hypertensive Arteriopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cerebral amyloid angiopathy: Patient with cerebral amyloid angiopathy
  Interventions: Other: None, pure observational study
- Hypertensive arteriopathy: Patients with hypertensive arteriopathy
  Interventions: Other: None, pure observational study

INTERVENTIONS:
Other: None, pure observational study — None, pure observational study

SUMMARY:
White matter hyperintensities (WMH) are one of the small vessel disease-related MRI characteristics of both cerebral amyloid angiopathy (CAA) and hypertensive arteriopathy (HA). WMH tend to show a peri-basal ganglia pattern in HA, whereas a multiple subcortical spots pattern can be observed in CAA. Periventricular WMH (PVWMH) have been reported to be posterior predominant using a semiautomated segmentation method and logarithmic transformation, not used in daily clinical practice. In these studies including CAA patients, patients initially presented with haemorrhage-related symptoms. In another study analysing PVWMH and cerebral amyloid evidence in patients with mild cognitive impairment, frontal PVWMH burden was associated with high uptake on florbetapir-PET whereas parietal and occipital PVWMH burden was associated with low CSF-amyloid-beta.

The aim of this study is the descriptive comparative analysis of the distribution of PVWMH between CAA and HA patients with radiological tools available in daily practice.

ELIGIBILITY:
Inclusion Criteria:

CAA and HA patients, managed at Nîmes University Hospital between January 2015 and March 2022.

Exclusion Criteria:

CAA and HA patients, treated at the CHU of Nîmes between January 2015 and March 2022, not objecting to the use of their health data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CAA and HA patients, managed at Nîmes University Hospital between January 2015 and March 2022
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Distribution of PVWMH | Base line, Day 0
  Maximal distance between the outer PVWMH border and the border of the lateral ventricle (on the axis oriented at 90° to the border of the ventricle)
Distribution of PVWMH - total PVWMH extent. | Base line, Day 0
  The sum of the PVWMH measurements around the four ventricles horns (i.e. bilateral anterior and posteriors horns) resulted in total PVWMH extent.
Corpus callosum (CC) WMH | Base line, Day 0
  Distance between the border of the third ventricle and the outer border of the WMH on the rostro-caudal axis, resulting in anterior and posterior CC-PVWMH extent measurements.
Corpus callosum (CC) WMH - total CC-PVWMH extent. | Base line, Day 0
  The sum of the anterior and posterior CC-PVWMH measurements resulted in the total CC-PVWMH extent.
Ratios | base line, day 0
  Calcul of posterior/anterior ratios for both the PVWMH and CC-PVWMH
Anterior PVWMH | Base line, Day 0
  Comparison of anterior PVWMH between CAA group and HA group.
Posterior PVWMH | Base line, Day 0
  Comparison of posterior PVWMH between CAA group and HA group.
Total PVWMH | Base line, Day 0
  Comparison of total PVWMH between CAA group and HA group.
Posterior/anterior PVWMH ratio | Base line, Day 0
  Comparison of the posterior/anterior PVWMH ratio between CAA and HA groups.
anterior CC-PVWMH | Base line, Day 0
  Comparison of anterior CC-PVWMH between CAA group and HA group.
Posterior CC-PVWMH | Base line, Day 0
  Comparison of posterior CC-PVWMH between CAA group and HA group.
Total PVWMH and posterior/anterior CC-PVWMH ratio | Base line, Day 0
  Comparison of total PVWMH and posterior/anterior CC-PVWMH ratio between CAA group and HA group.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Deasy L, Laurent-Chabalier S, Wacongne A, Parvu T, Mura T, Thouvenot E, Renard D. Diagnostic Accuracy of Posterior/Anterior Periventricular WMH Ratio to Differentiate CAA From Hypertensive Arteriopathy. Stroke. 2024 Aug;55(8):2086-2093. doi: 10.1161/STROKEAHA.123.046379. Epub 2024 Jun 26. PMID 38920025